CLINICAL TRIAL: NCT00181168
Title: Utility of Recombinant Human Thyrotropin (rTSH) PET-CT Fusion Scanning to Identify Residual Well-differentiated Epithelial Thyroid Cancer
Brief Title: Recombinant Thyrotropin PET-CT Fusion Scanning in Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Gustave Roussy, Cancer Campus, Grand Paris (Other); M.D. Anderson Cancer Center (Other); Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: THYR01105ORP; JHM IRB #1 (Other: Johns Hopkins University)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Thyroid Cancer
Keywords: thyroid cancer; PET scan; recombinant thyrotropin; thyroglobulin; Thyroid cancer, differentiated epithelial
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Thyrotropin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Euthyroid Group (Experimental): Euthyroid Group: Subjects received rhTSH to prepare for radioiodine therapy.
  Interventions: Drug: Euthyroid Group
- Hypothyroid Group (No Intervention): Hypothyroid Group: Thyroid hormone treatment was withheld before radioiodine therapy.

INTERVENTIONS:
Drug: Euthyroid Group — Euthyroid Group: Received rhTSH to prepare for radioiodine therapy.
  Other Names: Recombinant Human TSH (rhTSH)
  Arms: Euthyroid Group

SUMMARY:
The purpose of this study is to determine [for patients with previously treated well-differentiated thyroid cancer and evidence of residual disease based on serum thyroglobulin (Tg) level] whether positron emission tomography-computed tomography (PET-CT) fusion scanning performed after recombinant thyroid-stimulating hormone (TSH) (rTSH, thyrotropin alfa for injection) will be more sensitive for the detection of disease sites than PET-CT scanning without rTSH. The study will also determine if this information will significantly alter the therapeutic approach in some patients.

DETAILED DESCRIPTION:
PET/CT was performed before (basal PET) and 24 - 48 h after rhTSH administration (rhTSH-PET) in 63 patients (52 papillary and 11 follicular thyroid cancers). Images were blindly analyzed by two readers. The proposed treatment plan was prospectively assessed before basal PET, after basal PET, and again after rhTSH-PET.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged ≥ 18 years) with history of treated well-differentiated epithelial thyroid carcinoma (papillary, follicular or Hurthle cell), for which total or near total thyroidectomy plus postoperative radioiodine remnant ablation with 131-I has either been performed or found to be unnecessary by radioiodine imaging after TSH stimulation.
* Serum thyroglobulin (Tg) concentration ≥ 10 ng/mL (in the absence of interfering Tg autoantibodies).
* No findings of a "qualifying" radioiodine whole body scan that are sufficient to localize the disease suspected on the basis of the serum Tg.
* Inconclusive disease localization despite clinical assessment, cervical sonography, CT or magnetic resonance (MR) of the chest, and when appropriate other imaging and biopsy procedures. Patients must have no more than three foci of known or suspected extra-cervical metastasis.
* Must be in stable medical condition.
* Must be able to fully understand the protocol and be compliant with instructions.

Exclusion Criteria:

* Diabetes mellitus, due to interference with fluorodeoxyglucose (FDG) PET scanning.
* Claustrophobia, inability to lay supine, or other factors preventing cooperation with scanning procedures.
* Withdrawal of thyroid hormone or rTSH administration within the preceding month.
* Presence of circulating Tg autoantibodies interfering with serum Tg measurement.
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2001-03; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul W Ladenson, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (2):
  - Johns Hopkins Division of Endocrinology & Metabolism, Baltimore, Maryland
  - M.D. Anderson Cancer Center, Houston, Texas
- Institute Gustave Roussy, Paris, France

REFERENCES:
- [Background] Chin BB, Patel P, Cohade C, Ewertz M, Wahl R, Ladenson P. Recombinant human thyrotropin stimulation of fluoro-D-glucose positron emission tomography uptake in well-differentiated thyroid carcinoma. J Clin Endocrinol Metab. 2004 Jan;89(1):91-5. doi: 10.1210/jc.2003-031027. PMID 14715833
- [Result] Pacini F, Ladenson PW, Schlumberger M, Driedger A, Luster M, Kloos RT, Sherman S, Haugen B, Corone C, Molinaro E, Elisei R, Ceccarelli C, Pinchera A, Wahl RL, Leboulleux S, Ricard M, Yoo J, Busaidy NL, Delpassand E, Hanscheid H, Felbinger R, Lassmann M, Reiners C. Radioiodine ablation of thyroid remnants after preparation with recombinant human thyrotropin in differentiated thyroid carcinoma: results of an international, randomized, controlled study. J Clin Endocrinol Metab. 2006 Mar;91(3):926-32. doi: 10.1210/jc.2005-1651. Epub 2005 Dec 29. PMID 16384850
- [Result] Leboulleux S, Schroeder PR, Busaidy NL, Auperin A, Corone C, Jacene HA, Ewertz ME, Bournaud C, Wahl RL, Sherman SI, Ladenson PW, Schlumberger M. Assessment of the incremental value of recombinant thyrotropin stimulation before 2-[18F]-Fluoro-2-deoxy-D-glucose positron emission tomography/computed tomography imaging to localize residual differentiated thyroid cancer. J Clin Endocrinol Metab. 2009 Apr;94(4):1310-6. doi: 10.1210/jc.2008-1747. Epub 2009 Jan 21. PMID 19158200

RESULTS

PARTICIPANT FLOW:
Groups:
- Euthyroid Group: Subjects received rhTSH to prepare for radioiodine therapy
- Hypothyroid Group: Thyroid hormone treatment was withheld before radioiodine therapy.
Period: Overall Study
Arm/Group | Euthyroid Group | Hypothyroid Group
Started | 30 | 33
Completed | 30 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Euthyroid Group: Adults (age >18 years) with a history of treated well-differentiated epithelial thyroid carcinoma (papillary, follicular, or Hürthle cell), for which total or near total thyroidectomy plus postoperative radioiodine remnant ablation with 131-I has either been performed or found to be unnecessary by radioiodine imaging after TSH stimulation.
  Subjects received rhTSH to prepare for radioiodine therapy
- Hypothyroid Group: Adults (age >18 years) with a history of treated well-differentiated epithelial thyroid carcinoma (papillary, follicular, or Hürthle cell), for which total or near total thyroidectomy plus postoperative radioiodine remnant ablation with 131-I has either been performed or found to be unnecessary by radioiodine imaging after TSH stimulation.
  Thyroid hormone treatment was withheld before radioiodine therapy.
- Total: Total of all reporting groups
Arm/Group | Euthyroid Group | Hypothyroid Group | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 33 | 63
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 50
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  France | 13 | 14 | 27
  United States | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: PET-CT Fusion Scanning Sensitivity
Description: PET/CT was performed before (basal PET) and 24-48 h after rhTSH administration (rhTSH-PET) in 63 patients (52 papillary and 11 follicular thyroid cancers). Images were blindly analyzed by two readers. The proposed treatment plan was prospectively assessed before basal PET, after basal PET, and again after rhTSH-PET.
Time Frame: 21 Days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Euthyroid Group | Hypothyroid Group
Number analyzed (Participants) | 30 | 33
percentage of participants | 49 [36 to 62] | 54 [41 to 67]

2. Secondary Outcome: Increased Fluorodeoxyglucose (FDG) PET Standardized Uptake Value (SUV) After rTSH Specificity
Time Frame: 21 Days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | Euthyroid Group | Hypothyroid Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/33
Other Adverse Events (participants affected / at risk) | 0/30 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No